CLINICAL TRIAL: NCT03940872
Title: Development and Validation of a Diagnosis Questionnaire of Primary Parkinsonian Pain: the 3 PDQ Primary Parkinsonian Pain Diagnostic Questionnaire
Brief Title: Primary Parkinsonian Pain Diagnostic Questionnaire: Development and Validation of This Questionnaire
Acronym: 3PDQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC 31/18/0034
Record Dates: First submitted 2019-04-25; First posted 2019-05-07 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Parkinsonian central pain; Diagnosis; Primary Parkinsonian Pain Diagnostic Questionnaire
MeSH Terms: conditions — Parkinson Disease; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3PDQ self-questionnaire validation (Experimental): 200 patients will be included for this step in 10 French Parkinson expert centers.
  Interventions: Diagnostic Test: Self-questionnaire 3PDQ

INTERVENTIONS:
Diagnostic Test: Self-questionnaire 3PDQ — Visit 1 : - The patient will have to complete the 3PDQ self-questionnaire. - The investigator will conduct an interrogation and a neurological examination in order to ask or not the diagnosis of parkinsonian primary pain, without knowing the result of the 3PDQ.
  Visit 2 : - The patient will have to complete the 3PDQ self-questionnaire.
  - An investigator, obligatorily different from the investigator of the visit 1, will conduct to the same interrogation and the same neurological examination in order to ask or not the diagnosis of parkinsonian primary pain, without knowing the result of the 3PDQ.
  Visits 1 and 2 can be made on the same day. In this case the patient will fill the 3PDQ self questionnaire only once.

SUMMARY:
Development and validation of a diagnosis questionnaire of parkinsonian primary pain: the "Primary Parkinsonian Pain Diagnostic Questionnaire" (3PDQ)

DETAILED DESCRIPTION:
The aim of this study is to develop and validate a French self-questionnaire to diagnose parkinsonian primary : the "Primary Parkinsonian Pain Diagnostic Questionnaire" (3PDQ). It will allow clinicians to distinguish this pain from the other pain of the parkinsonian patient (whether or not related to Parkinson's disease).

The development and validation of the 3PDQ self-questionnaire will take place in 3 sequential steps:

1. design of the self-questionnaire
2. appearance validity study
3. validation of the self-questionnaire

Participants :

Appearance validity study: 40 painful parkinsonian patients Validation study: 200 painful parkinsonian patients (10 patients per item)

Duration of the study :

Duration of the inclusion period:

* Appearance validity study : 6 months
* Validity study : 20 months

Duration of participation for each patient:

* Appearance validity study : about 30 min
* Validity study : 3 days maximum Total duration of the study: (with results analysis): 3 years

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson Disease (PD)
* Patients who have chronic pain (for at least 3months) moderate to severe (intensity ≥ 4/10 on visual analogue scale from 0 to 10) specific or unspecific to PD
* Patients who have one type of pain or different type of pain: in this case, patients should suffered from one predominant pain and be able to identify it
* Patients who have stable analgesic medication during the study
* Patients who understand and speak fluently French
* Patients with health insurance
* Patients who signed the written informed consent form

Exclusion Criteria:

* Patients with severe depression according to Diagnostic and Statistical Manual (DSM) V criteria
* Analgesic medication modified recently (less than 1month)
* Patients with psycho-actives substances or alcohol abused
* Patients with cognitive impairment (MoCA score < 25)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Primary Parkinsonian Pain Questionnaire (3PDQ questionnaire) | 4 months
  Develop and validate a French self-questionnaire to diagnose parkinsonian primary pain, this symptom questionnaire will be called 3PDQ for Primary Parkinsonian Pain Questionnaire. This questionnaire present 5 items: Location of the most embarrassing pain, Characteristics of pain, if the pain is associated in the same area with one or more of the symptoms, by what is the pain caused or increased, what criteria does the pain correspond to.
  It is sufficient for each item to check the corresponding boxes

CONTACTS AND LOCATIONS:
Overall Officials: Christine BREFEL COURBON, MCU PH, Principal Investigator — Service de Pharmacologie Clinique et Service de Neurologie B8
Locations (10):
- France (10):
  - Neurology service, Clermont-Ferrand
  - Neurology service, Lille
  - Neurology service, Lyon
  - Neurology service, Marseille
  - Neurology Service, Montpellier
  - Neurolgoy service, Nancy
  - Neurology service, Nantes
  - Neurology service, Rouen
  - Neurology service, Strasbourg
  - Neurology service, Toulouse